CLINICAL TRIAL: NCT06233903
Title: A Prospective Study Assessing the Relationship Between Expression of the Norepinephrine Transporter and 18F-mFBG PET Imaging Results in Neuroblastoma Tumor, Other Neural Crest Tumors, and Organs Innervated by the Sympathetic Nervous System
Brief Title: 18F-mFBG Expression in Neural Crest Tumors and Organs Innervated by the Sympathetic Nervous System
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Logistical considerations
Sponsor: Innervate Radiopharmaceuticals LLC (Formerly: Illumina Radiopharmaceuticals LLC) (Industry)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRP101-201
Record Dates: First submitted 2024-01-05; First posted 2024-01-31 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Neuroblastoma; Pheochromocytoma; Paraganglioma
MeSH Terms: conditions — Neuroblastoma; Pheochromocytoma; Paraganglioma | interventions — 3-fluorobenzylguanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neural crest tumors and sympathetically innervated organs undergoing tissue sampling (Experimental): All subjects who undergo histopathologically established diagnosis of neuroblastoma and a scheduled clinical biopsy or surgery procedure within 21 days after 18F-mFBG PET imaging procedure; or be scheduled to have a clinical biopsy or surgery procedure that will yield a tissue specimen from an adrenergically-innervated organ or a non-neuroblastoma neural crest tumor within 21 days after 18F-mFBG PET imaging.
  Interventions: Drug: 18F-mFBG

INTERVENTIONS:
Drug: 18F-mFBG — 18F-mFBG positron emission tomography with CT (PET/CT) or positron emission tomography with MRI (PET/MRI)
  Other Names: Florbenguane F-18

SUMMARY:
This is a prospective Phase 2 study being performed to document the relationship between 18F-mIBG positron emission tomography (PET) findings in subjects, and expression of the norepinephrine transporter. In addition to collecting safety data for the imaging agent, the study aims to:

* compare the findings against other catacholamine transporters
* evaluate the imaging results at different time points and in different organs
* assess the quality of images with lower doses
* compare the ability to detect neuroblastoma lesions against other imaging agents, and in other tumors

DETAILED DESCRIPTION:
This is a prospective, Phase 2, open-label study designed to assess the relationship of 18F- mFBG PET imaging findings and NET expression in neuroblastoma tumor (Cohort I) and adrenergically-innervated organs in non-tumor subjects or neural crest tumors other than neuroblastoma (e.g. pheochromocytoma/paraganglioma) (Cohort II). As the mechanism of cellular uptake of benzylguanidine compounds such as mFBG is predominantly via cell-surface NET, there should be a demonstrable relationship between level of NET expression, whether expressed on neuroblastoma tumor, other neural crest tumors, or organs innervated by sympathetic neurons, and 18F-mFBG PET results. Eligible participants will either have: histopathologically established diagnosis of neuroblastoma and a scheduled clinical biopsy or surgery procedure within 21 days after 18F-mFBG PET imaging procedure; or be scheduled to have a clinical biopsy or surgery procedure that will yield a tissue specimen from an adrenergically-innervated organ or a non-neuroblastoma neural crest tumor within 21 days after 18F-mFBG PET imaging. At least one tissue specimen must be expected to be suitable for analysis of NET expression. Every subject will be expected to have at least 1 suitable recent tissue specimen available for NET expression analysis.

Neuroblastoma subjects will also have undergone at least 1 exam with the current standard of care benzylguanidine imaging agent, 123I-mIBG, during the course of clinical care following the original diagnosis of neuroblastoma.

All subjects will undergo 18F-mFBG PET imaging using either clinical PET/CT or PET/MRI equipment. PET studies will be examined on-site by a board-certified nuclear medicine physician or a board-certified radiologist experienced in reading 123I-mIBG and PET scans to ensure technical image quality and information content.

ELIGIBILITY:
Inclusion Criteria:

I. Neuroblastoma subjects (Cohort I)

1. The subject has an established diagnosis of neuroblastoma based on unequivocal histopathology from tissue obtained at any time prior to enrollment in the trial.
2. Functional imaging (123I-mIBG or 18F-FDG) studies performed within 60 days prior to receiving investigational drug in the trial are available for retrieval and independent review.
3. The subject is scheduled to undergo an invasive procedure (surgery or biopsy) for diagnosis or therapy of neuroblastoma within 21 days after receiving investigational drug in the trial, with no therapy in the interval between 18F-mFBG imaging and surgery/biopsy.
4. Histology specimens from the biopsy or surgical procedure are expected to be available and suitable for NET expression analyses.

   II. Non-neuroblastoma subjects (Cohort II):
5. The subject is scheduled to undergo an invasive procedure (surgery or biopsy) to obtain tissue from an adrenergically-innervated organ or a neural crest tumor within 21 days after 18F-mFBG imaging.
6. Histology specimens from the biopsy or surgical procedure are expected to be available and suitable for NET expression analyses.

   III. All subjects:
7. The subject is able and willing to comply with study procedures and a signed and dated informed consent (supplemented by signed and dated assent from subjects age 7-17) is obtained from the subject and/or at least 1 parent/guardian.

Exclusion Criteria:

Study Population

- The population will consist of either: subjects with histopathologically confirmed diagnosis of neuroblastoma; or subjects with a clinical indication for biopsy or surgical sampling of an adrenergically-innervated organ or a non-neuroblastoma neural crest tumor.

Inclusion Criteria:

Subjects will be eligible for participation in the study only if they meet ALL of the following criteria:

I. Neuroblastoma subjects (Cohort I)

1. The subject has an established diagnosis of neuroblastoma based on unequivocal histopathology from tissue obtained at any time prior to enrollment in the trial.
2. Functional imaging (123I-mIBG or 18F-FDG) studies performed within 60 days prior to receiving investigational drug in the trial are available for retrieval and independent review.
3. The subject is scheduled to undergo an invasive procedure (surgery or biopsy) for diagnosis or therapy of neuroblastoma within 21 days after receiving investigational drug in the trial, with no therapy in the interval between 18F-mFBG imaging and surgery/biopsy.
4. Histology specimens from the biopsy or surgical procedure are expected to be available and suitable for NET expression analyses.

   II. Non-neuroblastoma subjects (Cohort II)
5. The subject is scheduled to undergo an invasive procedure (surgery or biopsy) to obtain tissue from an adrenergically-innervated organ or a neural crest tumor within 21 days after 18F-mFBG imaging.
6. Histology specimens from the biopsy or surgical procedure are expected to be available and suitable for NET expression analyses.

   III. All subjects
7. The subject is able and willing to comply with study procedures and a signed and dated informed consent (supplemented by signed and dated assent from subjects age 7-17) is obtained from the subject and/or at least 1 parent/guardian.

Exclusion Criteria:

Subjects will not be eligible for participation in the study if they meet ANY of the following criteria:

1. Previously enrolled in this study.
2. Unable to lie flat or remain still for approximately 30 minutes to allow performance of a PET scan.
3. The subject has a history or suspicion of significant allergic reaction or anaphylaxis to any components of the 18F-mFBG imaging agent.
4. The subject is pregnant, breast feeding, or menarchal and unwilling to use effective contraception during the study.
5. Uses medications that are known to interfere with uptake of NET-dependent agents

   (e.g., certain antidepressants and sympathomimetics) and these medications cannot be safely withheld 24 hours before study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Norepinephrine Transporter (NET) expression | Tissue sampling completed within 22 days of 18F-mFBG imaging
  Norepinephrine Transporter (NET) expression of the sampled lesion(s)
Quantitation of 18F-mFBG uptake in sampled tissue | Analysis completed within 30 days of 18F-mFBG imaging
  Standard Uptake Value (SUV) from PET images from specific anatomic regions sampled

SECONDARY OUTCOMES:
Comparison of results at 30 vs. 60 minutes | 30 days after completion of 18F-mFBG imaging (Day 0)
  To evaluate whether 18F-mFBG imaging at 30 min yields results equivalent to those at 60 min post-injection. All image data files and processed/reconstructed PET images will undergo blinding and randomization. 18F-mFBG images will be qualitatively examined by 3 independent readers with no knowledge of the clinical status of the subjects but with access to anatomic cross-sectional images (CT or MRI) acquired as part of the PET exam.
Quality implications of reduced administered 18F-mFBG activity | 30 days after completion of 18F-mFBG imaging (Day 0)
  To assess the image quality implications of reducing the administered activity of 18F-mFBG. All image data files and processed/reconstructed PET images will undergo blinding and randomization. 18F-mFBG images will be qualitatively examined by 3 independent readers with no knowledge of the clinical status of the subjects but with access to anatomic cross-sectional images (CT or MRI) acquired as part of the PET exam. On-site image assessments will be performed per standard practice for PET imaging at the investigational site. Data for the on-site interpretations will be collected.
Comparison of 18F-mFBG disease detection at 60 minutes | 30 days after completion of 18F-mFBG imaging (Day 0)
  To determine if 18F-mFBG imaging at 60 min detects more neuroblastoma lesions than 123I-mIBG or 18F-FDG imaging. All image data files and processed/reconstructed PET images will undergo blinding and randomization. 18F-mFBG images will be qualitatively examined by 3 independent readers with no knowledge of the clinical status of the subjects but with access to anatomic cross-sectional images (CT or MRI) acquired as part of the PET exam.
Occurrence of adverse events in subjects with neuroblastoma | Up to 24 hours after each administration of 18F-mFBG injection
  To collect safety data on 18F-mFBG

CONTACTS AND LOCATIONS:
Overall Officials: Alice Lee, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States